CLINICAL TRIAL: NCT03501316
Title: Immune Response After Periodontal Treatment
Brief Title: The Immune Response After Periodontal Treatment
Acronym: iRaPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Michael Paterson, Honorary Clinical Lecturer in Restorative Dentistry, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iRaPT Research Study
Record Dates: First submitted 2018-03-13; First posted 2018-04-18 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Periodontal Diseases
Keywords: Root Surface Debridement; Hand Instrumentation; Ultrasonic Instrumentation; Systemic; Immune; CRP
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Analysis: the effect of treatment group (Manual vs ultrasonic) on changes in CRP levels (and other secondary outcomes):
  * Appropriate generalised linear models
  * Binary logistic models (for dichotomous outcomes)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the patients and clinicians will remain blinded to the intervention until the intervention is carried out. Research personnel will remain blinded to specific patient allocation throughout the process through the means of patient barcodes. The key linking the barcodes to the patients will be available to the Chief Investigator. The intervention codes will only be available once the key analyses have taken place.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Instrumentation (Active Comparator): Root surface debridement using hand instruments.
  Interventions: Device: Hand Instrumentation Treatment
- Ultrasonic Instrumentation (Active Comparator): Root surface debridement using ultrasonic scaler.
  Interventions: Device: Ultrasonic Instrumentation Treatment

INTERVENTIONS:
Device: Hand Instrumentation Treatment — Provision of treatment for periodontal disease using hand instrumentation. Following this, data will be collected relating to various factors, principle of which being systemic immune response.
  Arms: Hand Instrumentation
Device: Ultrasonic Instrumentation Treatment — Provision of treatment for periodontal disease using ultrasonic instrumentation. Following this, data will be collected relating to various factors, principle of which being systemic immune response.
  Arms: Ultrasonic Instrumentation

SUMMARY:
Primary Objective:

To identify changes in systemic markers of inflammation following periodontal treatment, comparing two standard treatment modalities (hands scaling and ultrasonic scaling)

Secondary Objectives:

To investigate bacteraemia, composition and function of oral bacteria, treatment outcomes following periodontal treatment, patient and operator preferences, and treatment time comparing hand scaling and ultrasonic scaling.

DETAILED DESCRIPTION:
Effective root surface debridement (RSD) is essential for successful periodontal treatment. Myriad studies demonstrate that RSD may be carried out using hand or ulstrasonic instruments with equal efficacy. Locally, effective debridement results in reduced inflammation in the gingival tissues, ultimately preserving the dentition. Systemically, RSD results in an immediate inflammatory response with elevated C-reactive protein (CRP), and cytokines (e.g. interleukin-6 and Tumor Necrosis Factor) detectable in the serum. This systemic inflammation may relate to systemic dissemination of bacteria from the periodontal pockets into the circulation, during instrumentation. Bacteria are detectable in serum immediately after instrumentation. The incidence of the bacteraemia varies considerably between different studies, ranging from 13% of patients to 43% to 55%. These studies used different methods of instrumentation; Kinane et al used full mouth ultrasonic scale, Zhang et al used a mixture of hand and ultrasonic instruments, and Heimdahl et al used curettes only. Whilst tempting to speculate that ultrasonic instrumentation induces less bacteraemia than hand instrumentation, there is no direct comparison of the effect of ultrasonic instrumentation with hand instrumentation on post treatment systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written, informed consent to participate
* Men or women aged 18 years to 70 years inclusive
* Periodontal disease requiring treatment at Glasgow Dental Hospital

Exclusion Criteria:

* Known or suspected high risk for tuberculosis, hepatitis B or HIV infections
* Require interpreter/non English language written material to understand and provide, or any other reason for being unable to provide written, informed consent
* History of bleeding diathesis
* Females using contraceptive methods.
* Pregnant or lactacting females.
* Reported diagnosis of any systemic illnesses including cardiovascular, renal, and liver diseases.
* Any pharmacological treatment within 3 months before the beginning of periodontal treatment.
* Specialist Periodontal treatment in the previous 6 months.
* Patients who will not tolerate Ultrasonic instrumentation even with local anaesthesia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Serum CRP | 24 hours after treatment, day 7, day 90
  Changes in serum CRP.

SECONDARY OUTCOMES:
Microbiome | Pre treatment and 24 hours after treatment
  Microbiome analysis of plaque
Bacteraemia analysis | Day 1, day 7, day 90 post intervention
  Bacteraemia analysis
Inflammation analysis | Day 1, 7 and 90 post treatment
  Gingival Crevicular Fluid - cytokine measurements
Periodontal Probing depths | day 90
  Periodontal Probing depths
Immune analysis | day 1, 7 and 90 post treatment
  Serum antibody measurement
Periodontal loss of attachment | day 90
  Index to determine the amount of connective tissue loss sustained by each tooth within the oral cavity as a result of the progressive, destructive periodontal disease process.
Gingivitis Index | day 90
  Levels of gingivitis within the oral cavity as a percentage of all tooth surfaces
Plaque Index | day 90
  Levels of plaque within the oral cavity as a percentage of all tooth surfaces
Blood pressure | day 1, 7 and 90 post treatment
  Blood pressure measured in millimeters of mercury. Measured using standard blood pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Shauna Culshaw, Principal Investigator — University of Glasgow
Locations (1):
- Michael Paterson, Glasgow, Glasgow City, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share data

REFERENCES:
- [Background] Ioannou I, Dimitriadis N, Papadimitriou K, Sakellari D, Vouros I, Konstantinidis A. Hand instrumentation versus ultrasonic debridement in the treatment of chronic periodontitis: a randomized clinical and microbiological trial. J Clin Periodontol. 2009 Feb;36(2):132-41. doi: 10.1111/j.1600-051X.2008.01347.x. PMID 19207889
- [Background] Graziani F, Cei S, Orlandi M, Gennai S, Gabriele M, Filice N, Nisi M, D'Aiuto F. Acute-phase response following full-mouth versus quadrant non-surgical periodontal treatment: A randomized clinical trial. J Clin Periodontol. 2015 Sep;42(9):843-852. doi: 10.1111/jcpe.12451. Epub 2015 Oct 1. PMID 26309133
- [Background] Horliana AC, Chambrone L, Foz AM, Artese HP, Rabelo Mde S, Pannuti CM, Romito GA. Dissemination of periodontal pathogens in the bloodstream after periodontal procedures: a systematic review. PLoS One. 2014 May 28;9(5):e98271. doi: 10.1371/journal.pone.0098271. eCollection 2014. PMID 24870125
- [Background] Kinane DF, Riggio MP, Walker KF, MacKenzie D, Shearer B. Bacteraemia following periodontal procedures. J Clin Periodontol. 2005 Jul;32(7):708-13. doi: 10.1111/j.1600-051X.2005.00741.x. PMID 15966875
- [Background] Zhang W, Daly CG, Mitchell D, Curtis B. Incidence and magnitude of bacteraemia caused by flossing and by scaling and root planing. J Clin Periodontol. 2013 Jan;40(1):41-52. doi: 10.1111/jcpe.12029. Epub 2012 Nov 9. PMID 23137266
- [Background] Heimdahl A, Hall G, Hedberg M, Sandberg H, Soder PO, Tuner K, Nord CE. Detection and quantitation by lysis-filtration of bacteremia after different oral surgical procedures. J Clin Microbiol. 1990 Oct;28(10):2205-9. doi: 10.1128/jcm.28.10.2205-2209.1990. PMID 2229342

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03501316/Prot_SAP_000.pdf